CLINICAL TRIAL: NCT04241016
Title: A Randomised Controlled Study of Endoscopic Sinus Surgery for Recurrent Acute Rhinosinusitis
Brief Title: Endoscopic Sinus Surgery in Recurrent Acute Rhinosinusitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Oulu University Hospital (Other)
Collaborators: Tampere University Hospital (Other)
Responsible Party: Principal Investigator, Olli-Pekka Alho, MD, Professor of Otorhinolaryngology, Oulu University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01234
Record Dates: First submitted 2020-01-17; First posted 2020-01-27 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Maxillary Sinusitis; Sinusitis, Acute; Sinusitis
Keywords: adult; endoscopic sinus surgery
MeSH Terms: conditions — Maxillary Sinusitis; Sinusitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endoscopic sinus surgery (ESS) (Active Comparator): Endoscopic sinus surgery. Postoperative treatment consists of daily nasal douching, daily nasal steroid sprays, pain medication when necessary and at least one postoperative control visit including endoscopy two weeks after the operation. Additionally medical treatment including nasal corticosteroids, nasal douching and other allergy medication as necessary.
  Interventions: Procedure: Endoscopic sinus surgery (ESS)
- Control (No Intervention): Conservative treatment including nasal corticosteroids, nasal douching and other allergy medication as necessary.

INTERVENTIONS:
Procedure: Endoscopic sinus surgery (ESS) — Uncinectomy, middle meatal antrostomy by enlarging the natural maxillary ostium and partial ethmoidectomy or septoplasty according to clinical evaluation of the operator.
  Arms: Endoscopic sinus surgery (ESS)

SUMMARY:
The aim of this study is to find out if endoscopic sinus surgery improves the quality of life in patients suffering from recurrent acute rhinosinusitis. Our main outcome is the difference between the average change in disease-specific SNOT-22 quality of life questionnaire scores (from baseline to 5-6 months follow-up) between the intervention and the control groups.

DETAILED DESCRIPTION:
This is a randomized controlled trial. Patients suffering from recurrent acute sinusitis episodes will be randomly allocated to two groups: intervention group, where they will receive endoscopic sinus surgery in addition to medical treatment and control group, where they will receive mere medical treatment. Both groups will be followed-up for 5 to 6 months. At baseline and after 5 to 6 months, patients will answer the life quality questionnaires SNOT-22 and RAND 36-item Health Survey. The numbers of sinusitis episodes, medical appointments for respiratory symptoms, use of medications, numbers of days lost from work or studies and numbers of days with various respiratory and adverse symptoms will be recorded with patient diaries. The potential serious adverse events (e.g. cerebrospinal fluid leak, orbital complications) related to surgery will be collected from the medical records.

ELIGIBILITY:
Inclusion Criteria:

* At least 3 acute sinusitis episodes during previous 6 months or 4 acute sinusitis episodes during previous 12 months or at least 2 episodes per year for 3 consecutive years
* Episodes must last less than 4 weeks and be diagnosed and treated as acute rhinosinusitis by a physician
* Episode symptoms include nasal discharge, nasal congestion, hyposmia and facial pressure or pain and the episodes have to be severe enough for the patient to seek medical help and for daily life to be significantly disturbed
* Patients must have failed a three-month conservative therapy (medication for possible allergies, nasal corticosteroids and douching and courses of antibiotics as necessary)

Exclusion Criteria:

* Age under 18 years,
* Immunodeficiency or immunosuppression
* Pregnancy,
* Previous illness making same-day surgery unfeasible
* Ongoing antibiotic treatment for other reasons,
* Primary complaint of nasal septal deviation and
* Chronic rhinosinusitis with or without nasal polyposis
* Symptoms for over 12 weeks and/or Lund-Mackay score over 8 in paranasal sinus CBCT scanning

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Sinonasal Outcome Test-22 score | 5-6 months
  Difference between the mean disease-specific Sinonasal Outcome Test 22 (SNOT-22) change scores (from baseline to 5-6 months) of ESS and control group. SNOT-22 summary scores vary between 0 and 110 with higher values indicating poorer quality of life.

SECONDARY OUTCOMES:
36-Item Short Form Survey (SF-36, RAND) score | 5-6 months
  Difference between the mean generic RAND-36 domains change scores (from baseline to 5-6 months) of ESS and control group. RAND-36 instrument produces eight individual values between 0 and 100 (one for each domain), with higher scores indicating better quality of life.
Difference in proportions of patients benefiting | 5-6 months
  Difference in proportions of patients benefiting clinically significantly from the treatment in ESS and control group (Minimum important change in SNOT-22 score)
Difference in numbers of sinusitis episodes | 5-6 months
  Difference in the numbers of sinusitis episodes between the ESS and control groups.
Difference in numbers of medical visits | 5-6 months
  Difference in the numbers of medical visits between the ESS and control groups.
Difference in numbers of antimicrobial treatments | 5-6 months
  Difference in the numbers of antimicrobial treatments between the ESS and control groups.
Difference in numbers of days lost from work or studies | 5-6 months
  Difference in the numbers of days lost from work or studies between the ESS and control groups.
Difference in numbers of days with nasal obstruction | 5-6 months
  Difference in the numbers of days with nasal obstruction between the ESS and control groups.
Difference in numbers of days with nasal discharge | 5-6 months
  Difference in the numbers of days with nasal discharge between the ESS and control groups.
Difference in numbers of days with facial pain or pressure | 5-6 months
  Difference in the numbers of days with facial pain or pressure between the ESS and control groups.
Difference in numbers of days with nasal pain | 5-6 months
  Difference in the numbers of days with nasal pain between the ESS and control groups.
Difference in numbers of days with nasal hemorrhage | 5-6 months
  Difference in the numbers of days with nasal hemorrhage between the ESS and control groups.
Difference of numbers of days with fever | 5-6 months
  Difference in the numbers of days with fever (>37.5 Celsius) between the ESS and control groups.
Adverse effects - postoperative synechia formation | 5-6 months
  Frequency of postoperative synechia formations in the ESS group
Adverse effects - postoperative infection | 5-6 months
  Frequency of postoperative infections in the ESS group
Adverse effects - postoperative orbital complication | 5-6 months
  Frequency of postoperative orbital complications in the ESS group
Adverse effects - postoperative intracranial complication | 5-6 months
  Frequency of postoperative intracranial complications in the ESS group

CONTACTS AND LOCATIONS:
Overall Officials: Olli-Pekka Alho, MD, PhD, Principal Investigator — Oulu University Hospital
Locations (2):
- Finland (2):
  - Oulu University Hospital, Oulu
  - Tampere University Hospital, Tampere

REFERENCES:
- [Derived] Kaski HM, Alakarppa A, Lantto U, Laajala A, Tokola P, Penna T, Ohtonen P, Alho OP. Endoscopic sinus surgery (ESS) to change quality of life for adults with recurrent rhinosinusitis: study protocol for a randomized controlled trial. Trials. 2021 Sep 8;22(1):606. doi: 10.1186/s13063-021-05576-z. PMID 34496924

DOCUMENTS (1):
  • Statistical Analysis Plan (2020-09-04): https://cdn.clinicaltrials.gov/large-docs/16/NCT04241016/SAP_000.pdf